CLINICAL TRIAL: NCT05819203
Title: Efficacy and Safety of Healsea® Babykids in the Treatment of Acute Infectious Rhinitis Symptoms in Children
Brief Title: BАbykids Spray In Common Cold
Acronym: BASICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lallemand Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LPH-2202
Record Dates: First submitted 2023-03-09; First posted 2023-04-19 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-04

CONDITIONS: Common Cold; Rhinitis Viral
Keywords: nasal spray; supplemented isotonic saline solution; infectious rhinitis; children
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial double blind
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigational device and the comparator were indistinguishable. The comparator (isotonic nasal spray) used the same technology and the same packaging than Healsea Babykids. A white label with regulatory mentions for clinical investigations was stuck on the vial A white label with regulatory mentions was sticked on a white cardboard box used as secondary packaging. The IFUs (Bulgarian version) was included in the secondary packaging (on one face, Healsea Babykids, on the other face Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healsea Babykids (Experimental): Healsea® Babykids, nasal spray indistinguishable from the comparator. Subjects have to spray 2 puffs in each nostril 2 times per day with a minimum of 7-day-treatment period (14 intakes ) up to 10 days (20 intakes ).
  Interventions: Device: Healsea Babykids
- Placebo (Placebo Comparator): The comparator is a saline isotonic nasal spray considered as inert Placebo i.e., neutral for the nasal mucosa.
  Subjects have to spray 2 puffs in each nostril 2 times per day with a minimum of 7-day-treatment period (14 intakes ) up to 10 days (20 intakes ).
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Healsea Babykids — 7-day-treatment period (14 intakes ) up to 10 days (20 intakes) .
  Arms: Healsea Babykids
Device: Placebo — 7-day-treatment period (14 intakes ) up to 10 days (20 intakes) .
  Arms: Placebo

SUMMARY:
The purpose of this post market clinical investigation is to demonstrate that Healsea® Babykids alleviates symptoms of the acute rhinitis phase with better efficacy than isotonic saline solution used as Placebo in children above 2 years.

DETAILED DESCRIPTION:
Healsea® Babykids is an isotonic saline solution based nasal spray supplemented with a natural Symbiofilm® extract (0.04%) isolated from marine bacteria. Symbiofilm® has in vitro antibiofilm activity and protects in vitro human nasal epithelial cells viability after Rhinovirus, Adenovirus, coronavirus OC43 and flu infection.

Healsea® Babykids is a nasal spray indicated in children above 2 years to clean and moisten the nose during colds and rhinitis.

The common cold is an acute viral infection of the upper respiratory tract, involving, to variable degrees, sneezing, nasal congestion and discharge (rhinorrhea), sore throat, cough, low-grade fever, headache, and malaise. Acute viral rhinitis is generally self-limiting. In children where the illness is not self-limiting and extends beyond 7-10 days, many agree that a bacterial infection is likely. Bacterial over infections and progression to a chronic state are favoured by the formation of biofilms, which facilitate bacterial growth and persistence as well as reducing antibiotic efficacy.

The aim of this study is to demonstrate that Healsea® Babykids alleviates symptoms of the acute rhinitis phase with better efficacy than isotonic saline solution used as Placebo.

The study comprises 2 parts:

- Part 1 (Day 1-Day 11): treatment of the acute phase

• with Healsea® Babykids, 2 puffs in each nostril 2 times per day with a minimum of 7-day-treatment period (14 intakes of Healsea® Babykids) up to 10 days (20 intakes of the investigational device).

or • with isotonic nasal spray (Placebo), 2 puffs in each nostril 2 times per day with a minimum of 7-day-treatment period (14 intakes of Placebo) up to 10 days (20 intakes of the investigational device).

- Part 2 (up to Day 15/Day 18): follow-up phase.

The study comprises two visits:

* Visit 1 (V1) at Day 1
* End of study visit (Visit 2, V2) between Day 15 and Day 18

ELIGIBILITY:
Inclusion Criteria:

* 1. Male/Female subjects >2 and ≤6-year-old
* 2. Acute infectious rhinitis/rhinosinusitis for ≤48h before trial entry
* 3. Patient presenting with fever ≥ 37.5 °C at screening
* 4. Subjects with nasal congestion (blocked / stuffy nose) rated at least as moderate on the Acute Rhinitis Symptoms Severity Questionnaire, based on evaluation by the investigator
* 5. Subjects showing at least moderate grade for at least one of the following additional signs of acute rhinitis: runny nose, nasal crust (dry mucus), sneezing and cough
* 6. Written consent obtained from parent/legal guardians

Exclusion Criteria:

* 1. Known hypersensitivity/allergy to any component of the test device
* 2. Medical history that is considered by the investigator as a reason for non-inclusion,
* 3. Severe nasal septum deviation or other condition that could cause nasal obstruction such as the presence of nasal polyps
* 4. History of nasal or sinus surgery that in the opinion of the investigator may influence symptom scores
* 5. Antibiotic intake within 2 weeks before screening
* 6. Systemic corticosteroids within 4 weeks before screening
* 7. Chronic decongestant use
* 8. Recent (within the previous 2 days) intake of a common cold medicine that in the opinion of the investigator may influence ARSSQ score at screening (NSAID, nasal decongestants, cough medicines)

Ages: 25 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rada MARKOVA, MD, Principal Investigator — Medical Center, Sofia
Locations (3):
- Bulgaria (3):
  - Medical center, Plovdiv
  - Medical center, Sofia
  - Medical center, Vratsa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Passioti M, Maggina P, Megremis S, Papadopoulos NG. The common cold: potential for future prevention or cure. Curr Allergy Asthma Rep. 2014 Feb;14(2):413. doi: 10.1007/s11882-013-0413-5. PMID 24415465
- [Result] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Result] Heikkinen T, Jarvinen A. The common cold. Lancet. 2003 Jan 4;361(9351):51-9. doi: 10.1016/S0140-6736(03)12162-9. PMID 12517470
- [Result] Principi N, Esposito S. Nasal Irrigation: An Imprecisely Defined Medical Procedure. Int J Environ Res Public Health. 2017 May 11;14(5):516. doi: 10.3390/ijerph14050516. PMID 28492494

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The comparator is a saline isotonic nasal spray considered as inert Placebo i.e., neutral for the nasal mucosa.
  Subjects have to spray 2 puffs in each nostril 2 times per day with a minimum of 7-day-treatment period (14 intakes ) up to 10 days (20 intakes ).
  Placebo: 7-day-treatment period (14 intakes ) up to 10 days (20 intakes) .
Period: Overall Study
Arm/Group | Healsea Babykids | Placebo
Started | 100 | 100
Completed | 98 | 98
Not Completed | 2 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healsea Babykids | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.9 (1.1) | 4.0 (1.2) | 4.0 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 52 | 51 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Curve (AUC) of the Global Score of the Acute Rhinitis Symptoms Severity Questionnaire (ARSSQ) During First 10 Days of Symptoms - Full Analysis Set (FAS)
Description: ARSSQ is a non-validated customized questionnaire. It includes 10 items assessing symptoms (questions 2 to 7), functional impairments (8 to 10), and global severity (question 1). Each item is scored from 0 (not present/no impact/ not sick) to 3 (severe, severe impact and very sick) for symptoms, functional impairment and global severity respectively. The questionnaire is to be completed in a diary once daily in the evening.
  The minimum ARSSQ score is zero (0) and the maximum ARSSQ score is thirty (30).
Time Frame: From Day 1 to Day 10
Population: FAS: all the subjects from the Safety Population and with at least one post-baseline efficacy data
Measure: Mean (Standard Deviation); unit: score on a scale*day
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
score on a scale*day | 78.1 (28.9) | 93.6 (28.9)
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Comparison of the means of AUC on global score or ARSSQ during the first 10 days of the study between both groups; Test type: Superiority; p = 0.0013, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Duration of Each Cold Symptom (Questions 2 to 7 of the ARSSQ) in Both Groups
Description: For each separate symptom, the duration is defined as the number of days between Day 1 and the first day the parent/legal guardian reports the patient not having this symptom ("Not present") for 2 consecutive days.
  Duration may be censored at Visit 2.
Time Frame: Through study completion, up to Day 18
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
Number of days | 6.92 (2.14) | 7.61 (2.05)
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Comparison of the mean duration of common cold during the study between both groups; Test type: Superiority; p = 0.0209, Cox survival regression and p Wald

3. Secondary Outcome: Duration of Quality-of-life Impairment (Questions 8 to 10 of the ARSSQ).
Description: as for outcome 2
Time Frame: Through study completion, up to Day 18
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Duration in Days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
Duration in Days | 6.46 (1.92) | 7.03 (1.97)
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Comparison of the mean duration of impact of common cold on quality of life during the study between both groups; Test type: Superiority; p = 0.0399, Cox survival regression and p Wald

4. Secondary Outcome: Cumulative Number of Days of Concomitant Treatments Use That May Affect Common Cold Symptoms (Antibiotics, Antipyretics, Systemic or Local Mucolytics, Decongestants, Antitussives, Systemic and Topical Corticosteroids)
Description: Concomitant treatments use (antibiotics, antipyretics, systemic or local mucolytics, decongestants, antitussives, systemic and topical corticosteroids) will be reported in the paper diary by parents/legal guardians throughout the study, validated by the investigator at the end of the study visit before being reported in the e-CRF.
Time Frame: Through study completion, up to Day 18
Population: Full Analysis Set
Measure: Number; unit: number of days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
number of days | 317 | 389
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Test type: Superiority; p = 0.0015, Poisson regression

5. Secondary Outcome: Cumulative Number of Days of Antibiotics Intake
Description: Antibiotics use will be reported in the paper diary by parents/legal guardians throughout the study, validated by the investigator at the end of the study visit before being reported in the e-CRF.
Time Frame: through study completion , up to day 18
Population: Full Analysis Set
Measure: Number; unit: number of days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
number of days | 108 | 127
Statistical Analysis 1: Comparison: Healsea Babykids; Test type: Superiority; p > 0.05, Poisson regression — not significant

6. Secondary Outcome: Cumulative Number of Days of Antipyretics Intake
Description: Antipyretics use will be reported in the paper diary by parents/legal guardians throughout the study, validated by the investigator at the end of the study visit before being reported in the e-CRF.
Time Frame: through study completion, up to day 18
Population: Full Analysis Set
Measure: Number; unit: number of days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
number of days | 62 | 86
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Test type: Superiority; p = 0.0029, Poisson regression

7. Secondary Outcome: Cumulative Number of Days of Mucolytics Intake
Description: Mucolytics use will be reported in the paper diary by parents/legal guardians throughout the study, validated by the investigator at the end of the study visit before being reported in the e-CRF.
Time Frame: Through study completion , up to day 18
Population: Full Analysis Set
Measure: Number; unit: number of days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
number of days | 44 | 85
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Test type: Superiority; p = 0.0006, Poisson regression

8. Secondary Outcome: Cumulative Number of Days of Decongestants Use
Description: Decongestants use will be reported in the paper diary by parents/legal guardians throughout the study, validated by the investigator at the end of the study visit before being reported in the e-CRF.
Time Frame: through study completion, up to day 18
Population: Full Analysis Set
Measure: Number; unit: number of days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
number of days | 149 | 220
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Test type: Superiority; p = 0.0513, Poisson regression

9. Secondary Outcome: Cumulative Number of Days of Antitussives Use
Description: Antitussives use will be reported in the paper diary by parents/legal guardians throughout the study, validated by the investigator at the end of the study visit before being reported in the e-CRF.
Time Frame: through study completion, up to day 18
Population: Full Analysis Set
Measure: Number; unit: number of days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
number of days | 23 | 18
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Test type: Superiority; p = 0.0789, Poisson regression

10. Secondary Outcome: Cumulative Number of Days of Systemic and Topical Corticosteroids Use
Description: Systemic and topical corticosteroids use will be reported in the paper diary by parents/legal guardians throughout the study, validated by the investigator at the end of the study visit before being reported in the e-CRF.
Time Frame: Through study completion, up to day 18
Population: Full Analysis Set
Measure: Number; unit: number of days
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 100 | 100
number of days | 25 | 66
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Test type: Superiority; p < 0.0001, Poisson regression

11. Primary Outcome: The Area Under the Curve (AUC) of the Global Score of the Acute Rhinitis Symptoms Severity Questionnaire (ARSSQ) During First 10 Days of Symptoms - Per Protocol Set (PP)
Description: as for outcome 1
Time Frame: From Day 1 to Day 10
Population: PP: efficacy population based on the FAS for subjects without major protocol deviation
Measure: Mean (Standard Deviation); unit: score on a scale*day
Arm/Group | Healsea Babykids | Placebo
Number analyzed (Participants) | 62 | 62
score on a scale*day | 80.5 (28.2) | 96 (29.5)
Statistical Analysis 1: Comparison: Healsea Babykids vs Placebo; Test type: Superiority — Comparison of the means of AUC on global score or ARSSQ during the first 10 days of the study between both groups; p = 0.0034, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the intervention through the study completion , up to day 18
Description: Reporting of adverse events and of incidents (Incident: any malfunction or deterioration in the characteristics or performance of a device made available on the market, including use-error due to ergonomic features, as well as any inadequacy in the information supplied by the manufacturer and any undesirable side-effect).
Arm/Group | Healsea Babykids | Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 11/100 | 14/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healsea Babykids (N=100) | Placebo (N=100)
tonsillitis (Infections and infestations) | 3 (3) | 5 (5)
otitis media acute (Infections and infestations) | 0 (0) | 2 (2)
Scarlet fever (Infections and infestations) | 1 (1) | 1 (1)
bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 0 (0) | 1 (1)
laryngitis (Infections and infestations) | 1 (1) | 0 (0)
pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
inner ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Adverse possibly related to the investigational device, ie incident reported to the competent authority per regulation EU 745/2017 , not rated as serious and did not lead to study /device discontinuation
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Adverse possibly related to the investigational device, ie incident reported to the competent authority per regulation EU 745/2017 , not rated as serious and did not lead to study /device discontinuation
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Adverse possibly related to the investigational device, ie incident reported to the competent authority per regulation EU 745/2017 , not rated as serious and did not lead to study /device discontinuation

LIMITATIONS AND CAVEATS:
In the absence of validated questionnaire assessing the severity and functional impact of an acute infectious rhinitis in young children, we used a customized non validated questionnaire, the ARSSQ (Acute Rhinitis Symptoms Severity Questionnaire).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05819203/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT05819203/SAP_001.pdf